CLINICAL TRIAL: NCT04095819
Title: Pilot Study to Evaluate Safety of and Efficacy of Middle Meningeal Artery (MMA) Embolization Compared to Traditional Surgical Strategies to Treat Chronic Subdural Hematomas (cSDH)
Brief Title: Middle Meningeal Artery (MMA) Embolization Compared to Traditional Surgical Strategies to Treat Chronic Subdural Hematomas (cSDH)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Atlantic Health System (Other)
Responsible Party: Principal Investigator, Ronald Benitez, MD, Director of Endovascular Surgery, Atlantic Health System
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AtlanticHS
Record Dates: First submitted 2019-09-09; First posted 2019-09-19 (Actual); Last update posted 2019-09-19 (Actual); Status verified 2019-09

CONDITIONS: Chronic Subdural Hematoma
MeSH Terms: conditions — Hematoma, Subdural, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Middle Meningeal Artery Embolization (Experimental): Middle Meningeal Artery Embolization
  Interventions: Procedure: Middle Meningeal Artery procedure
- Traditional Surgery (Active Comparator): Craniotomy/Burr hole
  Interventions: Procedure: Traditional Surgery

INTERVENTIONS:
Procedure: Middle Meningeal Artery procedure — Seal off the blood supply to the middle meningeal artery to prevent growth of the Subdural Hematoma
  Arms: Middle Meningeal Artery Embolization
Procedure: Traditional Surgery — Drainage of Subdural Hematoma using Craniotomy or Burr Hole
  Arms: Traditional Surgery

SUMMARY:
Chronic Subdural Hematoma (cSDH) is a common hematologic problem particularly in older patients. The purpose of this study is to evaluate the safety and efficacy of middle meningeal artery (MMA) embolization compared to traditional surgical strategies for patients presenting with chronic subdural hematoma (cSDH). Although MMA embolization is minimally-invasive procedure that is routinely used for the treatment of tumors or vascular formations (1), this study investigates the use of an established procedure for a new disease state.

DETAILED DESCRIPTION:
The purpose of the research study is to evaluate the safety and efficacy of a new, less-invasive procedure to treat chronic subdural hematoma (cSDH). A subdural hematoma occurs when blood collects on the brain's surface beneath the skull. Subdural hematomas can be life-threatening. They usually result from a head injury. This study will compare the new procedure to conventional surgical treatment of chronic subdural hematoma (cSDH). The new procedure is called middle meningeal artery embolization (MMA).

Current or conventional treatment of chronic subdural hematoma (cSDH) involves surgery (burr hole drainage and craniotomy) to access and remove the cause of the bleeding that is causing the subdural hematoma.

The new procedure, MMA embolization, involves guiding a catheter that is inserted into a blood vessel to the area of the brain that is supplying blood to the subdural hematoma. Particles or a special type of glue will be released to stop the bleeding that is causing the subdural hematoma. This technique has been used to treat other brain conditions, for example, (to treat tumors or malformation of blood vessels).

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Participant or Surrogate must be English speaking
* Subjects must have a diagnosis of chronic or acute-on subdural hematoma based on brain imaging, as documented by an
* One or more symptoms attributable to chronic SDH including headache cognitive impairment, gait instability, seizure, or mild focal neurologic deficit.
* In opinion of Investigator or the subject's referring physician, the subject has failed conservative management.

Exclusion Criteria:

* The Subdural hematoma is causing mass effect significant enough to cause marked or progressive neurologic impairment
* Any requirement for urgent surgical evacuation is necessary
* Life expectancy is less than 6 months in the opinion of the subject's primary physician
* Markedly tortuous vasculature precluding safe endovascular access, as assessed on angiogram
* Acute subdural hematomas
* Health insurance doesn't cover MMA embolization or performing Surgeon and follow up visits are considered out of network.
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-06-19 (Actual); Primary Completion 2022-04-19 (Estimated); Study Completion 2022-04-19 (Estimated)

PRIMARY OUTCOMES:
Change in size of SDH | 6 months
  Changes in size of SDH will be recorded in maximum diameter within 6 months.

SECONDARY OUTCOMES:
Change in Neurological status | 6 months
  Changes in Neurological status after the procedure and through study completion

CONTACTS AND LOCATIONS:
Locations (1):
- Overlook Medical Center, Summit, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fuentes AM, Khalid SI, Mehta AI. Predictors of Subsequent Intervention After Middle Meningeal Artery Embolization for Treatment of Subdural Hematoma: A Nationwide Analysis. Neurosurgery. 2023 Jan 1;92(1):144-149. doi: 10.1227/neu.0000000000002151. Epub 2022 Sep 21. PMID 36129273